CLINICAL TRIAL: NCT07091526
Title: Whether Controlling Serum Uric Acid (SUA) Can Benefit Postoperative Survival in Patients With Pancreatic Cancer
Brief Title: Whether Control of Serum Uric Acid (SUA) Improves Survival After Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: SUA-PC
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Serum Uric Acid
Keywords: Serum uric acid; Pancreatic cancer; Pancreaticoduodenectomy; Distal pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High serum uric acid: The increase of after serum uric acid operation compared with that before operation is≥10% Normal levels serum uric acid are typically 178 to 360 μm (3 to 6.8 mg/dl).
  Interventions: Diagnostic Test: serum uric acid test
- Low serum uric acid: The increase of after serum uric acid operation compared with that before operation < 10% Normal serum uric acid levels are typically 178 to 360 μm (3 to 6.8 mg/dl).
  Interventions: Diagnostic Test: serum uric acid test

INTERVENTIONS:
Diagnostic Test: serum uric acid test — Detect the serum uric acid in blood sample

SUMMARY:
This retrospective study aims to analyze the impact of postoperative changes in serum uric acid (SUA) levels on the prognosis of patients undergoing pancreatic cancer resection.

DETAILED DESCRIPTION:
Serum uric acid is a risk factor for gallbladder cancer in men and has a strong effect on pancreatic cancer in women. It has also been shown that elevated intracellular serum uric acid can induce an inflammatory stress response, which may promote its transformation, while elevated extracellular serum uric acidy further stimulate tumor cell proliferation, migration, and survival, and promote the development of highly aggressive cancer. In this study, the changes of serum uric acid before and after surgery was used as a prognostic marker for the survival of pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed pancreatic cancer (primary)
* Patients who underwent Radical resection of pancreatic cancer（Pancreaticoduodenectomy or Distal pancreatectomy）
* The postoperative survival time was at least 6 weeks

Exclusion Criteria:

* No surgery was performed, or only palliative surgery/ biopsy was performed
* Patients who underwent emergency hemodialysis or plasma exchange after surgery
* History of gout or long-term urate-lowering therapy, such as allopurinol
* Patients are missing follow-up data
* Hydrochlorothiazide and furosemide were used
* Chronic kidney disease
* Oncolytic syndrome
* Hemolytic anemia
* Lead poisoning
* Hyperparathyroidism
* Hypothyroidism
* A tyrosinase inhibitor was used
* Patients with nonpancreatic primary tumors
* Pregnant or postpartum women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radical pancreatic cancer resection patients
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-5 years
  Overall survival was defined as the time from diagnosis to death.

SECONDARY OUTCOMES:
Recurrence-free survival | 3-5 years
  Recurrence-free survival is the length of time from either the date of diagnosis or the start of therapy for a disease to the date of the first loco-regional or systemic recurrence.
Cost of hospitalization | 3 months
  The cost of the first hospitalization from admission to discharge.
Length of hospital stay | 3 months
  The first day of hospitalization for the first admission to the last day of discharge.
Pancreatic fistula | 3 months
  Whether or not pancreatic-intestinal anastomotic leakage occurred at the time of the first hospitalization.
Biliary fistula | 3 months
  Whether or not a biliary-intestinal anastomotic leak occurred at the time of the first hospitalization.
Bleeding | 3 months
  Whether or not there was bleeding after the first inpatient surgery.
Abdominal cavity infection | 3 months
  Whether or not there was an abdominal infection after the first inpatient surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D. Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang CF, Huang JJ, Mi NN, Lin YY, He QS, Lu YW, Yue P, Bai B, Zhang JD, Zhang C, Cai T, Fu WK, Gao L, Li X, Yuan JQ, Meng WB. Associations between serum uric acid and hepatobiliary-pancreatic cancer: A cohort study. World J Gastroenterol. 2020 Nov 28;26(44):7061-7075. doi: 10.3748/wjg.v26.i44.7061. PMID 33311950
- [Background] Fini MA, Elias A, Johnson RJ, Wright RM. Contribution of uric acid to cancer risk, recurrence, and mortality. Clin Transl Med. 2012 Aug 15;1(1):16. doi: 10.1186/2001-1326-1-16. PMID 23369448